CLINICAL TRIAL: NCT01084434
Title: Double-blind, Placebo Controlled Randomized Parallel Study to Determine the Effects of Pre-pro and Synbiotic Administration on the Immune Response to Influenza Vaccination and Faecal Microbiota in Healthy Adults
Brief Title: Probiotic, Prebiotic and Synbiotic Effect on Immunity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Reading (Other)
Responsible Party: Magdalena Baran, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F3168407
Record Dates: First submitted 2010-02-18; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-02

CONDITIONS: Dietary Intervention
MeSH Terms: interventions — Probiotics; Prebiotics; Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Probiotic group (Experimental): Group of 25 volunteers consuming probiotic product once a day for 7 weeks
  Interventions: Dietary Supplement: probiotic
- Prebiotic group (Experimental): Group of 25 volunteers consuming prebiotic product once a day for 7 weeks
  Interventions: Dietary Supplement: prebiotic
- Synbiotic group (Experimental): Group of 25 volunteers consuming synbiotic product once a day for 7 weeks.
  Interventions: Dietary Supplement: Synbiotic
- Placebo group (Placebo Comparator): Group of 25 volunteers consuming placebo product once a day for 7 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: probiotic — Bifidobacterium lactis HN019 10^9 CFU/day 1 sachet once a day for 7 weeks
  Other Names: HOWARU Bifidobacterium lactis
  Arms: Probiotic group
Dietary Supplement: prebiotic — Galactooligosaccharide 5.5 g/day 1 sachet once a day for 7 weeks
  Other Names: Bimuno
  Arms: Prebiotic group
Dietary Supplement: Synbiotic — (Bifidobacterium lactis 10^9 CFU + Galactooligosaccharide 5.5g) / day - 1 sachet once a day for 7 weeks
  Arms: Synbiotic group
Dietary Supplement: Placebo — Maltodextrin 5.5g/day - 1 sachet once a day for 7 weeks
  Arms: Placebo group

SUMMARY:
The aim of the study is to investigate the effect of dietary supplements such as probiotic, prebiotic and synbiotic on the immune response to influenza vaccination and faecal microbiota in adult healthy volunteers.

DETAILED DESCRIPTION:
Within recent times, influenza has become a major respiratory infection worldwide. The preventative vaccination reduces the severity of infection but ageing reduced its efficacy and it is only effective in 17-53% in elderly individuals. Thus, nutritionists and medical researchers are looking for opportunities to improve the immune response to influenza vaccine. Functional foods, such as probiotics, prebiotics and synbiotics, apart from other health benefits, may contribute towards immune protection.

Probiotics are beneficial bacteria, which are regarded as safe and serve health benefits to the host, while prebiotics are carbohydrates which by escaping digestion in the upper gastrointestinal tract may reach the colon and there serve as food for beneficial bacteria in the colon. When prebiotic used in combination with probiotic bacteria, it is called synbiotic, and it may improve survival and implantation of probiotic in the gut.

The human study will examine the immune response to vaccination and changes in faecal microbiota during administration of probiotic, prebiotic and synbiotic supplements. The study will be conducted between vaccinations seasons in 2010-2011 and recruit 100 healthy subjects aged 40-65years old. Participant will be given one of four different treatments over a 7 week period following 3 weeks of wash-out period. Treatments given include: a probiotic, a prebiotic, a synbiotic and a placebo. In the 3rd week of product consumption the participant will be given a flu jab. Specific antibody titre against the 3 viral strains composing the vaccine and total immunoglobulin concentration in the serum will be monitored during 2 and 4 weeks after vaccination. Faecal samples and saliva will be collected and analysed for changes in faecal microbial populations.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Age 40-65 years
* Body mass index 18.5-30 inclusive
* Good general health as determined by medical questionnaires
* Not vaccinated with the current seasonal influenza (2009) or swine flu vaccine

Exclusion Criteria:

* Evidence of physical or mental disease or planned major surgery, which might limit participation in or completion of the study
* History of drug misuse, including alcohol
* Allergy to the vaccine
* Asplenia and other acquired or congenital immunodeficiency
* Severe allergy such as asthma, hay-fever, dermatitis or being treated on these
* History of severe abnormal drug reaction
* Any autoimmune disease
* Diabetic (type 1 or type2)
* Food allergy manifested by gastrointestinal, skin, respiratory , neurological, anaphylaxis symptoms
* Lactose intolerance showed by clinical symptoms such as nausea, cramping, bloating, diarrhea and flatulence after consuming lactose containing dairy products (milk, yoghurt, butter, cheese, ice-cream, sour cream) or lactose non-dairy products ( whey, milk solids, modified milk ingredients)
* Participation in experimental drug trial within four weeks prior to study
* Participation in prebiotics or laxative trial within the previous three months
* Use of antibiotics within the previous six months
* Chronic constipation, diarrhoea or other chronic gastro-intestinal complaint
* Intake of other prebiotics or probiotics, drugs active on gastrointestinal motility, or a laxative of any class for four weeks prior to study
* Use of prescribed medication
* Regular use of aspirin or other anti-inflammatory drugs

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome would be a higher change in antibody levels in response to influenza vaccination compared to placebo group. | 2 and 4 weeks after vaccination

SECONDARY OUTCOMES:
The secondary outcome would be a change in faecal microbiota groups and a change in their metabolic activities. | at 0, 7 and 10 weeks on pro-, pre,synbiotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Magdalena Baran, MSc, Principal Investigator; Sofia Kolida, PhD, Principal Investigator
Locations (1):
- University of Reading, Food and Nutritional Sciences Department, Reading, Berkshire, United Kingdom